CLINICAL TRIAL: NCT07019220
Title: COBRA - Chemoablation for Low Grade Bladder Cancer: A Single Arm, Prospective, Open-label, Investigator-initiated Phase 2 Study
Brief Title: Chemoablation for Low-Grade Bladder Cancer
Acronym: COBRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ekaterina Laukhtina (Other)
Responsible Party: Sponsor-Investigator, Ekaterina Laukhtina, Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COBRA
Record Dates: First submitted 2025-06-04; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: Non-Muscle Invasive Bladder Cancer; Intravesical Therapy; Non-Surgical Treatment
MeSH Terms: conditions — Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with low-grade NMIBC (Experimental)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Intravesical installation

SUMMARY:
The goal of this single arm, prospective, open-label, investigator-initiated Phase 2 clinical trial is to evaluate the efficacy of intravesical chemoablation in patients with low grade bladder cancer.

DETAILED DESCRIPTION:
In this study, patients with histologically confirmed Ta low-grade bladder cancer will undergo chemoablation with gemcitabine (six weekly instillations). The study aims to evaluate the efficacy, safety, and tolerability of chemoablation.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of providing documented informed consent will be enrolled in this study
* Diagnosis of a recurrent tumor and a history of TaLG BCa or diagnosis of primary TaLG BCa histologically confirmed by cold cup biopsy at screening or within 8 weeks before screening
* On screening cystoscopy: Diameter of the largest lesion ≤15mm
* Number of lesions ≤5
* Cystoscopy with bladder diagram including number, site, size and appearance of the tumors with photo documentation
* Patient who has recurrence of and not other than TaLG NMIBC (low or intermediate EAU risk)
* NMIBC requiring treatment with transurethral resection of bladder tumors (TURBT)
* Negative voiding cytology for high grade (HG) disease within 8 weeks before Screening
* No lymph node metastasis or distant metastasis
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment. Female patients of childbearing potential must use adequate contraception during study period
* Willing and able to provide informed consent

Exclusion Criteria:

* Tumors that clinicians suspect to be HG
* Positive HG cytology according to Paris criteria
* Diameter of tumor >15 mm
* Number of lesions >5
* Any previous intravesical therapy within 1 year
* Previous HG NMIBC (within the last 3 years). It is allowed to include patients who had history of HG disease longer than 3 years ago.
* Past or current muscle invasive bladder cancer (i.e., T2, T3, T4) or metastatic UC
* History of upper tract urothelial carcinoma (UTUC)
* Clinically significant urethral stricture that would preclude passage of a urethral catheter
* History of neurogenic bladder; active urinary retention; any other condition that would prohibit normal voiding
* Evidence of active urinary tract infection (UTI) that in the Investigator's opinion cannot be treated and resolved prior to biopsy and/or administration of study treatment
* Patient refused to participate
* Known positive human immunodeficiency virus (HIV) test.
* Female patients who are pregnant/breastfeeding.
* Female patients of childbearing potential not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (cCR) | From the end of treatment (EOT) visit to the follow-up visits (1 and 3 months post-treatment).
  cCR defined as negative urine cytology and absence of macroscopic tumor at the cystoscopic evaluation

SECONDARY OUTCOMES:
Pathological complete response (pCR) | From the end of treatment visit (EOT) to the follow-up visits (1 and 3 months post-treatment).
  pCR defined as negative urine cytology, absence of macroscopic tumor at cystoscopic evaluation and confirmed by negative biopsy/TURB
Patient-reported Outcomes based on EORTC QLQ-NMIBC24 | Will be measured weekly during treatment period, at the end of treatment visit and follow-up visits (1 and 3 months post-treatment).
  The global health status/quality of life endpoint will be based on the scales of EORTC QLQ-NMIBC24 questionnaire.
Patient-reported Outcomes based on EORTC QLQ-C30 | Will be measured weekly during treatment period, at the end of treatment visit and follow-up visits (1 and 3 months post-treatment).
  The global health status/quality of life endpoint will be based on the scales of EORTC QLQ-C30 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shahrokh F. Shariat Prof. Dr., Professor, Principal Investigator — Department of Urology, Medical University of Viernna
Locations (1):
- Department of Urology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
The data collected in this study includes sensitive patient information related to medical history, treatment responses, and clinical outcomes. To protect patient confidentiality and comply with ethical guidelines and institutional policies, individual participant data will not be shared publicly

REFERENCES:
- [Background] Brausi MA, Gontero P, Altieri V, Colombo R, Conti I, Bono AV. Can gemcitabine instillation ablate solitary low-risk non-muscle-invasive bladder cancer? Results of a phase II marker lesion study. Urol Int. 2011;87(4):470-4. doi: 10.1159/000331727. Epub 2011 Nov 11. PMID 22086229
- [Background] Gardmark T, Carringer M, Beckman E, Malmstrom PU; Members of the Intravesical Gemcitabine Study Group. Randomized phase II marker lesion study evaluating effect of scheduling on response to intravesical gemcitabine in recurrent Stage Ta urothelial cell carcinoma of the bladder. Urology. 2005 Sep;66(3):527-30. doi: 10.1016/j.urology.2005.03.084. PMID 16140071
- [Background] Maffezzini M, Campodonico F, Canepa G, Capponi G, Fontana V. Short-schedule intravesical gemcitabine with ablative intent in recurrent Ta-T1, G1-G2, low- or intermediate-risk, transitional cell carcinoma of the bladder. Eur Urol. 2007 Apr;51(4):956-61. doi: 10.1016/j.eururo.2006.08.038. Epub 2006 Sep 20. PMID 17027141
- [Background] Campodonico F, Canepa G, Capponi G, Bozzo L, Maffezzini M. Intravesical gemcitabine in recurrent superficial bladder carcinoma: preliminary results on ablative efficacy and tolerability. Anticancer Res. 2005 May-Jun;25(3c):2381-4. PMID 16080464
- [Background] Serretta V, Galuffo A, Pavone C, Allegro R, Pavone-MacAluso M. Gemcitabine in intravesical treatment of Ta-T1 transitional cell carcinoma of bladder: Phase I-II study on marker lesions. Urology. 2005 Jan;65(1):65-9. doi: 10.1016/j.urology.2004.08.027. PMID 15667865
- [Background] Gontero P, Casetta G, Maso G, Sogni F, Pretti G, Zitella A, Frea B, Tizzani A. Phase II study to investigate the ablative efficacy of intravesical administration of gemcitabine in intermediate-risk superficial bladder cancer (SBC). Eur Urol. 2004 Sep;46(3):339-43. doi: 10.1016/j.eururo.2004.05.001. PMID 15306105